CLINICAL TRIAL: NCT05719701
Title: A Multi-center, Non-randomized, and Open-label Phase I/IIa Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of ICP-490 in Patients With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Evaluate the Safety, Tolerability, and Efficacy of ICP-490 in Patients With Relapsed and/or Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01101
Record Dates: First submitted 2023-01-10; First posted 2023-02-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Relapsed and/or Refractory Multiple Myeloma
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICP-490 (Experimental)
  Interventions: Drug: ICP-490
- ICP-490 in combination with Dexamethasone (Experimental)
  Interventions: Drug: ICP-490; Drug: Dexamethasone

INTERVENTIONS:
Drug: ICP-490 — Several dose groups of ICP-490 are planned for the dose exploration.
Drug: Dexamethasone — Oral Dexamethasone is administered on Days 1, 8, 15, and 22 of each 28-day cycle.
  Arms: ICP-490 in combination with Dexamethasone

SUMMARY:
This is a multi-center, non-randomized and open-label phase I/IIa clinical study to evaluate the safety, tolerability, and efficacy of ICP-490 in patients with relapsed and/or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 years old.
2. Diagnosed as relapsed and/or refractory multiple myeloma .The patient must have measurable diseases.Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-2.
3. Patients must have adequate organ function. Expected survival time ≥ 6 months.
4. All toxicities caused by prior anticancer therapy must have recovered to Grade ≤ 1 (based on CTCAE v5.0) except alopecia and fatigue.

Female patients of childbearing potential should have a negative blood pregnancy test result within 48 h prior to the first dose of investigational drug.

Exclusion Criteria:

1. Known active central nervous system (CNS) involvement or history of the disease, or clinical signs of multiple myeloma meningeal/spinal meningeal involvement.
2. Patients with solitary plasmacytoma; plasma cell leukemia (PCL) (active PCL or history of PCL); Waldenström's macroglobulinemia; POEMS syndrome or symptomatic amyloidosis.
3. Prior active or history of malignancies other than MM, occurring within 5 years prior to the first dose of investigational drug, with the exception of radically treated local curable cancers.
4. Uncontrolled or severe cardiovascular disorders.
5. Any active infection within 14 days prior to the first dose of investigational drug.
6. Patients with diseases restricted from participation as described in the protocol
7. Having undergone major surgery within 28 days prior to the first dose of investigational drug, or minor surgery within 2 weeks prior to the first dose. Any severe or uncontrolled systemic disease evaluated by investigatorthat may increase the risk associated with study participation and drug administration or affect the patient's ability to receive the investigational drug.
8. Patients who have received any other systemic treatment, anti-tumor traditional Chinese (herbal) medicine therapy , and any other investigational drug therapy for MM within 28 days or 5 half-lives of the drugs (whichever is shorter) prior to the first dose of investigational drug.
9. Patients who have received systemic treatment with corticosteroids or other immunosuppressive drugs within 14 days prior to the first dose of investigational drug.

   Subjects are allowed to use topical, ocular, intra-articular, intranasal, and inhaledcorticosteroid ; short-term use (≤ 7 days) of corticosteroid for prophylaxis (e.g., contrast agent allergy) or for the treatment of non-autoimmune diseases (e.g., delayed hypersensitivity reaction caused by contact allergens) is permitted.
10. Patients who have received medications or foods with strong inhibitory or inductive effects on cytochrome P450 CYP3A, and proton pump inhibitorswithin 2 weeks prior to the first dose of investigational drug, or are planning to receive them during the study.
11. Patients with a history of severe allergic reactions to IMIDs , or dexamethasone, or to any component contained in ICP-490 or dexamethasone formulation (CTCAE V5.0 Grade > 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Phase I : Incidence, type, and severity of adverse events (AEs) as judged according to NCI-CTCAE V5.0 | Through study completion, an average of 3 years
  AE refers to any adverse event occurring in subjects during clinical research period. The incidence and type of AEs will be evaluated and the severity will be judged according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version5.0.
Phase I : Incidence, type, and severity of dose-limiting toxicities (DLTs) | Through study completion, an average of 3 years
  The dose-limiting toxicity (DLT) assessed in the phase I dose exploration study is defined as AEs related to study treatment that meet the following criteria (according to the NCI CTCAE v5.0 criteria) and occur in Cycle 1.
Phase I : RP2Ds and/or MTDs | Through study completion, an average of 3 years
  Phase I is the dose exploration study of ICP-490 to preliminarily determine RP2Ds (probably more than one) and MTD (if applicable). MTD: The dose level corresponding to the dose group whose posterior probability of DLT incidence estimated by PAVA (pool adjacent violators algorithm) is closest to the target toxicity probability (25%).
Phase II : ORR (defined as sCR + CR + VGPR + PR) assessed according to IMWG criteria. | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | Through study completion, an average of 3 years
  Maximum concentration (Cmax) will be calculated through multiple plasma concentrations drawn from the patients after administration.
Time to maximum concentration (Tmax) | Through study completion, an average of 3 years
  Time to maximum concentration (Tmax) will be calculated through multiple plasma concentrations drawn from the patients after administration.
Half-life (T1/2) | Through study completion, an average of 3 years
  Half-life (T1/2) will be calculated through multiple plasma concentrations drawn from the patients after administration.
Area under the concentration-time curve (AUC0-∞ and AUC0-t) | Through study completion, an average of 3 years
  Area under the concentration-time curve (AUC0-∞ and AUC0-t) will be calculated through multiple plasma concentrations drawn from the patients after administration.
Apparent clearance (CL/F) | Through study completion, an average of 3 years
  Apparent clearance (CL/F) will be calculated through multiple plasma concentrations drawn from the patients after administration.
Apparent volume of distribution during terminal phase (Vz/F) | Through study completion, an average of 3 years
  Apparent volume of distribution during terminal phase (Vz/F) will be calculated through multiple plasma concentrations drawn from the patients after administration.
Steady-state PK parameters | Through study completion, an average of 3 years
  Steady-state PK parameters will be calculated through multiple plasma concentrations drawn from the patients after administration.
The overall response rate (ORR) assessed according to the International Myeloma Working Group (IMWG) criteria (ORR, defined as stringent complete response (sCR) + complete response (CR) + very good partial response (VGPR) + partial response (PR)) | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria.
Phase I & IIa : Complete response rate (CRR, defined as sCR + CR) assessed according to IMWG criteria | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria.
Phase I & IIa : Very good or better partial response rate assessed according to IMWG criteria (≥ VGPR rate, defined as VGPR + sCR + CR) | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria.
Phase I & IIa : Time to response (TTR) assessed according to IMWG criteria | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria
Phase I & IIa : Duration of response (DOR) assessed according to IMWG criteria | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria
Phase I & IIa : Progression-free survival (PFS) assessed according to IMWG criteria | Through study completion, an average of 3 years
  Disease response will be assessed according to the 2016 IMWG response criteria
Phase I & IIa : Overall survival (OS) | Through study completion, an average of 3 years
  The follow-up visits should be carried out every 12 weeks after the last dose via telephone or other methods to obtain the survival status information of patients.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hosptital, Zhengzhou, Henan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital，Zhejiang University School of Medicine, Hangzhou, Zhejiang